CLINICAL TRIAL: NCT02060318
Title: The Effect of Infliximab Therapy in Crohn Patients on Regulatory T-cells
Brief Title: Regulatory T-cells and Crohn's Disease
Acronym: CrohnReg
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ove Andersen, MD, PhD, Hvidovre University Hospital
Other Study IDs: H-1-2013-072; HVH-2013-028 (Registry Identifier: Datatilsynet)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Regulatory T-cells; Infliximab
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infliximab: 35 Crohn patients about to start Infliximab treatment, gives as i.v. injection of 5 mg/kg at baseline, after 2 weeks, 6 weeks, and then every 8th week.
  Interventions: Drug: Infliximab
- Healthy controls: 12 healthy controls without Crohn's Disease.

INTERVENTIONS:
Drug: Infliximab — The patients are included in the study when the decision to treat with Infliximab is already made. This study is observational, and all treatment and clinical follow-up are according to national guidelines.
  Groups: Infliximab

SUMMARY:
Aim: the main aim of this study is to investigate if immune cells (regulatory T-cells, Th17 cells and other immune cell types) or biomarkers can be used to predict the response or lack of response to treatment with Infliximab. If so, characteristics of the immune cells may also unveil the mechanisms behind lack of response to Infliximab.

Design: a prospective, observational study with three arms. In the treatment group, 35 patients with Crohn's disease about to start Infliximab-treatment are recruited. They have blood samples drawn at day 1 before first treatment, after 6 week, and again after 22 weeks of treatment. 12 healthy volunteers serve as a control group. Controls are only investigated once. All treatment and follow-up are according to national guidelines, and data from this study is not used by the clinicians.

Methods: the number of regulatory T-cells and pro-inflammatory T-cells (Th17 cells) is investigated using flow cytometry. From plasma and serum samples, various proteins (biomarkers), such as transforming growth factor beta (TGF-beta) and tumour necrosis factor alpha (TNF-alpha), are measured using immunoassays. Patient data (demographics and medical history) are extracted from various registries.

DETAILED DESCRIPTION:
Primary analyses: patient response to Infliximab treatment is quantified using Harvey Bradshaw Index, and the response is then related to the number of regulatory T-cells, Th17 cells, and biomarker levels at baseline. The exact cut-off for response vs. non-respons will be determined and validated once all data is collected by an assessor blinded for the flow cytometry results and biomarker levels.

Plan for missing data: for patients with missing Harvey Bradshaw Index, we will first try to re-create the score using the patient records (information on well-being, abdominal pain, diarrhea, fistulae/abscesses, and extra-intestinal Crohn manifestations). If this is not possible, an experienced clinician will rate the patient's Infliximab response based on all available patient record data, but blinded for flow cytometry results and biomarker levels.

ELIGIBILITY:
Infliximab group

Inclusion Criteria:

* Crohn's Disease
* Starting Infliximab treatment
* Patient at the gastrointestinal department at Hvidovre Hospital or Køge Sygehus
* Can understand and write Danish
* European ancestry

Exclusion Criteria:

* Not able to consent in an ethical manner (e.g. severe mental illness)
* Significant co-morbidity (e.g. cancer, HIV)
* Other immunological disease (e.g. psoriasis)
* Current treatment with biological agents

Healthy controls

Inclusion Criteria:

* No current disease
* No daily drug use
* Can understand and write Danish
* European ancestry

Exclusion Criteria:

* Not able to consent in an ethical manner (e.g. severe mental illness)
* Significant co-morbidity (e.g. cancer, HIV)
* Other immunological disease (e.g. psoriasis)
* Current treatment with biological agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the gastroenterology department at Hvidovre Hospital and Køge Sygehus are eligible for entry.
  Healthy controls are recruited by advitising at Hvidovre Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2016-03-07 (Actual); Study Completion 2016-03-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of regulatory T-cells at 6 weeks | Baseline, 6 weeks (plus/minus 1 week)
  The number of regulatory T-cells is measured in fresh blood by flow cytometry.
Change from baseline in number of regulatory T-cells at 22 weeks | Baseline, 22 weeks (plus/minus 1 week)
  The number of regulatory T-cells is measured in fresh blood by flow cytometry.

SECONDARY OUTCOMES:
Change from baseline in Harvey Bradshaw Index at 6 weeks | Baseline, 6 weeks (plus/minus 1 week)
  Harvey Bradshaw Index is a measure of Crohn's Disease severity.
Change from baseline in CD161 expression at 6 weeks | Baseline, 6 weeks (plus/minus 1 week)
  Cluster of differentiation 161 (CD161) is a T helper 17 cell (Th17)-marker, measured by flow cytometry of fresh blood samples.
Change from baseline in CD161 expression at 22 weeks | Baseline, 22 weeks (plus/minus 1 week)
  CD161 is a Th17-marker, measured by flow cytometry of fresh blood samples.
Change from baseline in cytokine levels at 6 weeks | Baseline, 6 weeks (plus/minus 1 week)
  We will measure IFN-gamma, IL-4, IL-6, IL-7, IL-10, IL-15, IL-17, and TNF-alpha by Luminex. TGF-beta, suPAR, and IL-15 will be measured by ELISA.
Change from baseline in cytokine levels at 22 weeks | Baseline, 22 weeks (plus/minus 1 week)
  We will measure IFN-gamma, IL-4, IL-6, IL-7, IL-10, IL-15, IL-17, and TNF-alpha by Luminex. TGF-beta, suPAR, and IL-15 will be measured by ELISA.
Change from baseline in Harvey Bradshaw Index at 22 weeks | Baseline, 22 weeks (plus/minus 1 week)
  Harvey Bradshaw Index is a measure of Crohn's Disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, MD, PhD, Principal Investigator — Hvidovre Hospital & University of Copenhagen
Locations (1):
- Hvidovre Hospital, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data sets will be made available on relevant requests and in accordance with journal guidelines when publishing results from this study.